CLINICAL TRIAL: NCT01732783
Title: Prospective Observational Cohort Study to Describe the Use of Vectibix® in Combination With Chemotherapy in Routine Clinical Practice for Patients With Wild-type RAS Metastatic Colorectal Cancer
Brief Title: Observational Study of Vectibix With Chemotherapy for Metastatic Colorectal Cancer Patients
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: 20120100
Record Dates: First submitted 2012-11-20; First posted 2012-11-26 (Estimated); Results first posted 2018-08-20 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Wild-type RAS Metastatic Colorectal Cancer
Keywords: Wild-type RAS; Metastatic Colorectal Cancer; Vectibix
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Panitumumab; Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Metastatic Colorectal Cancer: Participants with wild-type RAS metastatic colorectal cancer who were receiving panitumumab in combination with chemotherapy.
  Interventions: Other: Panitumumab + Chemotherapy

INTERVENTIONS:
Other: Panitumumab + Chemotherapy — Participants receiving panitumumab in combination with chemotherapy as prescribed by the treating physician prior to enrollment in this study and according to routine clinical practice for patients with wild-type RAS metastatic colorectal cancer.
  Other Names: Vectibix®

SUMMARY:
The primary objective was to describe the pattern of use of panitumumab (Vectibix®) in combination with chemotherapy in patients with wild-type rat sarcoma viral oncogene homolog (RAS) metastatic colorectal cancer (mCRC): as first-line treatment in combination with FOLFOX or FOLFIRI or second-line treatment in combination with FOLFIRI in patients who have received first-line fluoropyrimidine-based chemotherapy (excluding irinotecan).

ELIGIBILITY:
Inclusion Criteria

* Subject is ≥ 18 years of age at date of enrolment
* Histologically or cytologically confirmed carcinoma of colon or rectum
* Subject with metastatic carcinoma of colon or rectum
* Confirmed wild-type RAS status of tumour
* Subjects whose care will be managed primarily by the enrolling physician and/ or all records will be available
* Tumour assessment (ie, computed tomography [CT]/magnetic resonance imaging [MRI]) within 12 weeks (84 days) prior to first Vectibix® infusion.
* Subjects treated with at least one infusion of Vectibix® in combination with chemotherapy a maximum of 84 days before entering study: first-line in combination with FOLFOX (folinic acid, leucovorin, fluorouracil [5FU], oxaliplatin) or second-line in combination with FOLFIRI (folinic acid, leucovorin, 5FU, irinotecan) in subjects who have received first-line fluoropyrimidine-based chemotherapy (excluding irinotecan) for treatment of wild-type RAS mCRC per approved prescribing information
* Subject or subject's legally acceptable representative has provided informed consent (for countries where required per local regulations)
* Subjects treated with Vectibix® in accordance with the current version of the Summary of Product Characteristics (SmPC)

Exclusion Criteria

* Ongoing or planned concurrent participation in any clinical study involving Investigational Product that has not been approved by the European Medicines Agency for any indication
* Ongoing or planned concurrent participation in any clinical study where the dosing of Vectibix® is determined by the protocol (participation in clinical trials on an approved drug and observational trials are permitted but these cannot mandate how mCRC should be treated)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All treatment centres (inpatient and outpatient) with a focus on treating patients with mCRC. Centres will be selected to represent academic, oncology and specialist settings and to provide geographical diversity in France and Germany.
Sampling Method: Non-Probability Sample
Enrollment: 213 (Actual)
Dates: Start 2012-12-10 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2016-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in France and Germany between 10 December 2012 and 30 November 2016.
Groups:
- Panitumumab + FOLFOX First-line: Participants with metastatic colorectal cancer (mCRC) with tumor expressing wild-type RAS who received panitumumab in combination with FOLFOX as first-line treatment (FLFAS).
- Panitumumab + FOLFIRI Second-line: Participants with mCRC with tumor expressing wild-type RAS who received panitumumab in combination with FOLFIRI as second-line treatment and received first-line fluoropyrimidine-based chemotherapy (excluding irinotecan) (SLFAS).
- Panitumumab + FOLFIRI First-line: Participants with mCRC with tumor expressing wild-type RAS who received panitumumab in combination with FOLFIRI as first-line treatment (FLFFAS).
Period: Overall Study
Arm/Group | Panitumumab + FOLFOX First-line | Panitumumab + FOLFIRI Second-line | Panitumumab + FOLFIRI First-line
Started | 164 | 37 | 12
Completed | 29 (Completed 12-month observation period.) | 5 (Completed 12-month observation period.) | 2 (Completed 12-month observation period.)
Not Completed | 135 | 32 | 10
Not completed — Discontinued Panitumumab Treatment | 106 | 25 | 7
Not completed — Death | 13 | 4 | 1
Not completed — Lost to Follow-up | 7 | 1 | 1
Not completed — Administrative Decision | 8 | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Panitumumab + FOLFOX First-line | Panitumumab + FOLFIRI Second-line | Panitumumab + FOLFIRI First-line | Total
Number analyzed (Participants) | 164 | 37 | 12 | 213
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (9.6) | 65.8 (9.9) | 69.0 (7.6) | 65.2 (9.5)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 73 | 18 | 2 | 93
  ≥ 65 to < 75 years | 68 | 14 | 7 | 89
  ≥ 75 years | 23 | 5 | 3 | 31
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 13 | 5 | 70
  Male | 112 | 24 | 7 | 143
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — A scale to assess a patient's disease status. 0 = Fully active, able to carry out all pre-disease performance without restriction; 1 = Restricted in physically strenuous activity, ambulatory and able to carry out work of a light nature; 2 = Ambulatory and capable of all self-care, unable to carry out any work activities. Up and about > 50% of waking hours; 3 = Capable of only limited self-care, confined to bed or chair > 50% of waking hours; 4 = Completely disabled, confined to bed or chair; 5 = Dead.
  Participants
    0 - Fully active | 44 | 7 | 4 | 55
    1 - Restricted but ambulatory | 28 | 11 | 3 | 42
    2 - Ambulatory but unable to work | 8 | 2 | 0 | 10
    Missing | 84 | 17 | 5 | 106
Primary Colorectal Cancer Type [Count of Participants; unit: Participants]
  Colon, left of mid-line | 54 | 14 | 4 | 72
  Colon, right of mid-line | 41 | 8 | 7 | 56
  Colon | 3 | 2 | 0 | 5
  Rectum | 66 | 13 | 1 | 80
Metastatic Colorectal Cancer Status [Count of Participants; unit: Participants] — Synchronous colorectal neoplasias are defined as 2 or more primary tumors identified in the same patient and at the same time.
  Metachronous refers to lesions that appear after diagnosis of the primary lesion.
  Participants
    Synchronous | 115 | 20 | 5 | 140
    Metachronous | 39 | 14 | 7 | 60
    Missing | 9 | 2 | 0 | 11
    Unknown | 1 | 1 | 0 | 2
Metastatic Disease Lesion Sites [Number; unit: participants]
  Liver | 123 | 25 | 5 | 153
  Lung | 36 | 13 | 4 | 53
  Other | 56 | 11 | 4 | 71

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Panitumumab Infusions
Time Frame: 12 months
Measure: Median (Inter-Quartile Range); unit: infusions
Arm/Group | Panitumumab + FOLFOX First-line | Panitumumab + FOLFIRI Second-line | Panitumumab + FOLFIRI First-line
Number analyzed (Participants) | 164 | 37 | 12
infusions | 10.0 [6.0 to 16.0] | 10.0 [6.0 to 16.0] | 8.0 [4.0 to 15.5]

2. Primary Outcome: Cumulative Dose of Panitumumab
Time Frame: 12 months
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | Panitumumab + FOLFOX First-line | Panitumumab + FOLFIRI Second-line | Panitumumab + FOLFIRI First-line
Number analyzed (Participants) | 164 | 37 | 12
mg | 4262.5 [2311.5 to 6902.5] | 4000.0 [2400.0 to 6000.0] | 3782.5 [1772.5 to 5751.0]

3. Primary Outcome: Maximum Dose of Panitumumab
Time Frame: 12 months
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | Panitumumab + FOLFOX First-line | Panitumumab + FOLFIRI Second-line | Panitumumab + FOLFIRI First-line
Number analyzed (Participants) | 164 | 37 | 12
mg | 450.0 [380.0 to 520.0] | 420.0 [390.0 to 500.0] | 507.0 [424.0 to 590.0]

4. Primary Outcome: Duration of Panitumumab Exposure
Description: Duration of exposure is the time from the first to the last panitumumab infusion
Time Frame: 12 months
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Panitumumab + FOLFOX First-line | Panitumumab + FOLFIRI Second-line | Panitumumab + FOLFIRI First-line
Number analyzed (Participants) | 164 | 37 | 12
months | 5.339 [2.546 to 10.053] | 6.012 [2.464 to 8.246] | 5.339 [1.922 to 12.008]

5. Primary Outcome: Mean Interval Between Panitumumab Infusions
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Panitumumab + FOLFOX First-line | Panitumumab + FOLFIRI Second-line | Panitumumab + FOLFIRI First-line
Number analyzed (Participants) | 163 | 37 | 12
Participants
  > 0 to 7 days | 0 | 0 | 0
  > 7 to 14 days | 38 | 7 | 2
  > 14 to 21 days | 98 | 22 | 4
  > 21 to 28 days | 21 | 8 | 5
  > 28 days | 6 | 0 | 1

6. Primary Outcome: Percentage of Participants With at Least One Panitumumab Dose Reduction
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Panitumumab + FOLFOX First-line | Panitumumab + FOLFIRI Second-line | Panitumumab + FOLFIRI First-line
Number analyzed (Participants) | 164 | 37 | 12
percentage of participants | 36.6 [29.6 to 44.2] | 21.6 [11.4 to 37.2] | 50.0 [25.4 to 74.6]

7. Primary Outcome: Percentage of Participants With at Least One Panitumumab Dose Delay
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Panitumumab + FOLFOX First-line | Panitumumab + FOLFIRI Second-line | Panitumumab + FOLFIRI First-line
Number analyzed (Participants) | 164 | 37 | 12
percentage of participants | 42.7 [35.4 to 50.3] | 21.6 [11.4 to 37.2] | 41.7 [19.3 to 68.0]

8. Primary Outcome: Reasons for Discontinuation of Panitumumab
Time Frame: 12 months
Population: Participants who discontinued panitumumab while on study
Measure: Count of Participants; unit: Participants
Arm/Group | Panitumumab + FOLFOX First-line | Panitumumab + FOLFIRI Second-line | Panitumumab + FOLFIRI First-line
Number analyzed (Participants) | 138 | 34 | 8
Participants
  Disease progression | 35 | 12 | 3
  Physician or Oncologist decision | 30 | 7 | 0
  Planned surgical resection | 16 | 1 | 0
  Death | 12 | 3 | 1
  Adverse Drug Reaction (ADR) | 11 | 4 | 2
  Patient request to discontinue all treatment | 9 | 1 | 2
  Adverse event | 8 | 1 | 0
  Lost to follow-up | 6 | 1 | 0
  Other | 6 | 1 | 0
  Patient request to discontinue panitumumab | 5 | 3 | 0

9. Primary Outcome: Duration of Exposure of All Concomitant Chemotherapy
Description: Duration of exposure is the time from the first date to the last date of chemotherapy administration.
Time Frame: 12 months
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Panitumumab + FOLFOX First-line | Panitumumab + FOLFIRI Second-line | Panitumumab + FOLFIRI First-line
Number analyzed (Participants) | 164 | 37 | 12
months | 5.240 [2.595 to 8.969] | 5.092 [2.431 to 7.622] | 3.860 [1.889 to 9.413]

10. Primary Outcome: Percentage of Participants With at Least One Concomitant Chemotherapy Dose Reduction
Time Frame: 12 months
Measure: Number; unit: percentage of participants
Arm/Group | Panitumumab + FOLFOX First-line | Panitumumab + FOLFIRI Second-line | Panitumumab + FOLFIRI First-line
Number analyzed (Participants) | 164 | 37 | 12
percentage of participants | 43.3 | 24.3 | 58.3

11. Primary Outcome: Percentage of Participants With at Least One Concomitant Chemotherapy Dose Delay
Time Frame: 12 months
Measure: Number; unit: percentage of participants
Arm/Group | Panitumumab + FOLFOX First-line | Panitumumab + FOLFIRI Second-line | Panitumumab + FOLFIRI First-line
Number analyzed (Participants) | 164 | 37 | 12
percentage of participants | 29.3 | 29.7 | 33.3

12. Secondary Outcome: Number of Participants With at Least One Hospitalization
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Panitumumab + FOLFOX First-line | Panitumumab + FOLFIRI Second-line | Panitumumab + FOLFIRI First-line
Number analyzed (Participants) | 164 | 37 | 12
Participants | 163 | 37 | 12

13. Secondary Outcome: Types of Hospital Visit
Description: Participants may have had more than one type of hospital visit.
Time Frame: 12 months
Population: Participants with at least one hospital visit
Measure: Number; unit: participants
Arm/Group | Panitumumab + FOLFOX First-line | Panitumumab + FOLFIRI Second-line | Panitumumab + FOLFIRI First-line
Number analyzed (Participants) | 163 | 37 | 12
participants
  Outpatient | 157 | 35 | 12
  Inpatient | 75 | 12 | 6
  Emergency room | 11 | 1 | 0
  Day case | 6 | 2 | 0
  Other | 6 | 1 | 0

14. Secondary Outcome: Duration of Hospital Stay
Time Frame: 12 months
Population: Participants with at least one hospital visit
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Panitumumab + FOLFOX First-line | Panitumumab + FOLFIRI Second-line | Panitumumab + FOLFIRI First-line
Number analyzed (Participants) | 163 | 37 | 12
days | 40.0 [19.0 to 66.0] | 28.0 [19.0 to 43.0] | 24.5 [8.5 to 60.5]

15. Secondary Outcome: Reasons for Hospitalization
Description: Participants may have had more than one hospital visit and/or reason for a hospital visit.
Time Frame: 12 months
Population: Participants with at least one hospitalization
Measure: Number; unit: participants
Arm/Group | Panitumumab + FOLFOX First-line | Panitumumab + FOLFIRI Second-line | Panitumumab + FOLFIRI First-line
Number analyzed (Participants) | 163 | 37 | 12
participants
  mCRC related | 144 | 30 | 10
  Treatment-related | 88 | 16 | 9
  mCRC and treatment related | 74 | 14 | 7

16. Secondary Outcome: Percentage of Participants With an Overall Response
Description: Tumor response was assessed by the investigator using standard radiological imaging. Overall response is defined as a best tumor response of complete response or partial response according to Response Evaluation Criteria In Solid Tumours (RECIST).
Time Frame: 12 months
Population: Participants with tumor response data post-baseline
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Panitumumab + FOLFOX First-line | Panitumumab + FOLFIRI Second-line | Panitumumab + FOLFIRI First-line
Number analyzed (Participants) | 124 | 33 | 8
percentage of participants | 47.6 [38.5 to 56.7] | 33.3 [18.0 to 51.8] | 50.0 [15.7 to 84.3]

17. Secondary Outcome: Number of Participants With Resectability
Description: Resectability denotes whether a participant became resectable during the study.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Panitumumab + FOLFOX First-line | Panitumumab + FOLFIRI Second-line | Panitumumab + FOLFIRI First-line
Number analyzed (Participants) | 164 | 37 | 12
Participants
  Yes | 20 | 3 | 1
  No | 135 | 33 | 7
  Unknown | 9 | 1 | 4

18. Secondary Outcome: Number of Participants With Anti-cancer Treatment After Panitumumab Discontinuation
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Panitumumab + FOLFOX First-line | Panitumumab + FOLFIRI Second-line | Panitumumab + FOLFIRI First-line
Number analyzed (Participants) | 164 | 37 | 12
participants | 84 | 15 | 3

19. Secondary Outcome: Type of Post-Panitumumab Anti-cancer Treatment
Description: Participants may have received more than one type of anti-cancer treatment that was initiated after panitumumab discontinuation.
Time Frame: 12 months
Population: Participants who reported use of anti-cancer treatment after discontinuation of panitumumab
Measure: Number; unit: participants
Arm/Group | Panitumumab + FOLFOX First-line | Panitumumab + FOLFIRI Second-line | Panitumumab + FOLFIRI First-line
Number analyzed (Participants) | 84 | 15 | 3
participants
  Chemotherapy | 72 | 10 | 3
  Other | 10 | 2 | 0
  Radiotherapy | 5 | 0 | 1
  Targeted biologics | 5 | 3 | 1
  Other small molecules | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: From first dose of panitumumab until 30 days after last dose, or up to the 12 month end of study observation period, whichever occurred first; median reporting period was 6.3, 7.0, and 6.3 months for each group respectively.
Description: Only adverse reactions considered by the investigator to be related to panitumumab together with product complaints and other safety findings were collected in this observational study.
  Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Panitumumab + FOLFOX First-line | Panitumumab + FOLFIRI Second-line | Panitumumab + FOLFIRI First-line
All-Cause Mortality (participants affected / at risk) | 0/164 | 0/37 | 0/12
Serious Adverse Events (participants affected / at risk) | 10/164 | 0/37 | 0/12
Other Adverse Events (participants affected / at risk) | 101/164 | 25/37 | 8/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Panitumumab + FOLFOX First-line (N=164) | Panitumumab + FOLFIRI Second-line (N=37) | Panitumumab + FOLFIRI First-line (N=12)
Angina pectoris (Cardiac disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0
Inflammation of wound (Injury, poisoning and procedural complications) | 1 | 0 | 0
Eastern Cooperative Oncology Group performance status worsened (Investigations) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Dermatosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Collapse circulatory (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Panitumumab + FOLFOX First-line (N=164) | Panitumumab + FOLFIRI Second-line (N=37) | Panitumumab + FOLFIRI First-line (N=12)
Diarrhoea (Gastrointestinal disorders) | 7 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 1 | 1
Mucosal inflammation (General disorders) | 10 | 2 | 2
Conjunctivitis (Infections and infestations) | 2 | 3 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 10 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 7 | 3 | 0
Rash (Skin and subcutaneous tissue disorders) | 80 | 21 | 6
Skin fissures (Skin and subcutaneous tissue disorders) | 8 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.